CLINICAL TRIAL: NCT06429540
Title: Evaluation of Post Extraction Hard Tissue Alteration Following Ridge Preservation Using Partially Demineralized Dentin Block Versus Xenograft in the Esthetic Zone: A Randomized Controlled Clinical Trial
Brief Title: Post Extraction Changes Following Ridge Preservation Using Partially Demineralized Dentin Block Versus Xenograft
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Danah Tayseer Al Ghothani, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12224PER6-3-1
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Socket Preservation
Keywords: L-PRF; Xenograft; Collagen membrane; Dentin block; Partially demineralized dentin block; Socket preservation; Liquid fibrinogen
MeSH Terms: interventions — Transplantation, Heterologous

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Clinical Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partially Demineralized Dentin Block (Experimental): The Partially Demineralized Dentin Block will be prepared using the Tooth Transformer device to grind the extracted tooth and partially demineralize it. Leukocyte-Platelet Rich Fibrin (L-PRF) and liquid fibrinogen will then be added to create a block graft.
  Interventions: Biological: Partially Demineralized Dentin Block
- Xenograft (Active Comparator): The Xenograft procedure will involve filling the socket with deproteinized bovine bone mineral, followed by the placement of a collagen membrane to cover the socket
  Interventions: Biological: Xenograft

INTERVENTIONS:
Biological: Partially Demineralized Dentin Block — The extracted tooth will be dried using air, then ground and partially demineralized with the Tooth Transformer device following the manufacturer's protocol. Dentin particles will be obtained with dimensions of 400-800 μm. The partially demineralized dentin will then be prepared by cutting the Leukocyte-Platelet Rich Fibrin (L-PRF) membranes into small pieces and mixing them with the dentin particles. Liquid fibrinogen will be added to the homogeneous mixture. Within a few minutes, the fibrinogen will convert into fibrin primarily from the activated blood platelets in the chopped L-PRF membranes. This process will effectively trap the biomaterial and the L-PRF pieces, forming the "dentin block". After that, the sockets will be carefully packed with the dentin block and it will be covered with L-PRF membrane. To ensure stability and prevent displacement, the wounds will be secured using non-resorbable sutures.
  Arms: Partially Demineralized Dentin Block
Biological: Xenograft — In the control group using the Xenograft, the same extraction and socket debridement procedure will be performed. Following that, the extraction socket will be thoroughly filled with deproteinized bovine bone mineral, and a collagen membrane will be employed to cover the socket. The membrane will be shaped to extend 2-3 mm beyond the margins of the extraction socket and positioned just beneath the marginal mucosa. To ensure its stability, a cross-suture will be performed, securing the membrane in place.
  Arms: Xenograft

SUMMARY:
The aim of this study is to clinically and radiographically evaluate the dimensional changes of hard tissue after using Partially Demineralized Dentin Block versus Xenograft in the esthetic zone.

The main question: In patients with unrestorable teeth, will the use of partially demineralized Dentin Block be more effective than Xenograft in preserving vertical and horizontal ridge dimensions?

After enrollment, a thorough preoperative assessment, including history taking, clinical, and radiographic examinations, will be conducted.

Initial therapy includes periodontal treatment (phase 1 therapy) followed by random assignment to one of two treatment groups: ridge preservation using Partially Demineralized Dentin Block or Xenograft.

Both groups will undergo atraumatic extraction.

For the test group, an autogenous partially demineralized dentin graft will be prepared, involving tooth cleaning, grinding, and partial demineralization with the Tooth Transformer device, followed by Leukocyte-Platelet Rich Fibrin (L-PRF) membrane and liquid fibrinogen preparation. The L-PRF membranes will be cut, mixed with dentin particles, and combined with liquid fibrinogen to form a compact graft. The block will be placed inside the socket and covered by an L-PRF membrane and secured with a cross-suture.

In the control group, Xenograft will be used, and the socket filled with deproteinized bovine bone mineral, covered with a collagen membrane, and secured with a cross-suture.

After a healing period of 6 months, at the time of implant placement, a biopsy will be taken using a trephine bur.

DETAILED DESCRIPTION:
Objective of the study: The aim of this study is to evaluate post extraction hard tissue changes following ridge preservation using Partially Demineralized Dentin Block versus Xenograft in the esthetic zone.

Research Procedure: Patients will be selected from the outpatient clinic of the Oral Medicine and Periodontology Department, Faculty of Dentistry, Cairo University.

General operative procedures: Patients who fulfill the inclusion criteria will be enrolled. The nature of the study will be explained to each patient, as well as the importance of compliance with pre- and post-operative instructions and follow-up visits.

Preoperative preparation: A thorough preoperative assessment of all patients will be carried out, including history taking, clinical examination, and radiographic examination.

History: Each patient will be interviewed to obtain a comprehensive history.

Clinical examination: Proper intraoral examination will be done to evaluate the following parameters for the tooth of interest: 1) Restorability of the tooth. 2) Periodontal condition of the tooth to be extracted and the adjacent teeth.

Radiographic examination:

1. Periapical radiographs will be done to rule out the presence of any periapical infection and evaluate the presence of caries or periodontal disease in the adjacent teeth.
2. In cases that meet the inclusion criteria, cone beam computed tomography (CBCT) will be taken at three time points: before the surgery, immediately after socket preservation, and after 6 months. The CBCT before the surgery will be used to assess the type of socket, while the baseline CBCT immediately after socket preservation will be used to evaluate the horizontal ridge width at 1, 3, and 5 mm below the most coronal aspect of the crest, and buccal and palatal ridge height. The CBCT taken after 6 months will serve to superimpose the two scans and assess long-term changes.

Initial Therapy: The initial therapy will consist of periodontal treatment (phase I therapy) including supragingival scaling, subgingival debridement if needed, adjustment of faulty restorations, and polishing. Mechanical plaque control instructions for each patient include brushing and interdental cleaning techniques.

Patients will be randomly assigned to one of the treatment groups:

* Test Group: Ridge preservation using Partially Demineralized Dentin Block in the esthetic zone.
* Control Group: Ridge preservation using Xenograft in the esthetic zone.

Surgical Procedure:

Atraumatic extraction:

* The patient will rinse with 0.12% Chlorhexidine (Hexitol, ADCO Pharma Co, Egypt).
* The operator will administer 4% articaine hydrochloride with 1:100,000 epinephrine (Septodent Co. for Pharmaceuticals, France).
* Flapless and atraumatic tooth extraction will be initiated by making an intrasulcular incision using a 15c blade.
* Next, a periotome will be used to sever the periodontal ligament (PDL) fibers, followed by the use of a straight elevator and extraction forceps for the extraction process.

In the test group, the autogenous partially demineralized dentin graft will be prepared as follows: A high-speed fine finishing stone and saline irrigation will be used to clean the tooth and remove any decay, restoration, or foreign materials. The tooth will be rinsed twice in phosphate buffered saline. The tooth will be dried using air, then ground and partially demineralized with the Tooth Transformer device following the manufacturer's protocol. Dentin particles will be obtained with dimensions of 400 - 800 μm.

Dentin block preparation: During the preparation of partially demineralized dentin, Leukocyte-Platelet Rich Fibrin (L-PRF) membranes will also be prepared. Vacutainer tubes without anticoagulant (red cap, glass coating) will be used to collect four 10-cc blood samples, which will then be immediately centrifuged at 2700 rpm for 12 minutes using the IntraSpin centrifuge (IntraLock, Florida, USA). Additionally, two extra blood samples will be collected in 9-cc non-coated vacutainer tubes without anticoagulants (white cap). These samples will be centrifuged at 2700 rpm for 3 minutes. The resulting yellow fluid (liquid fibrinogen) at the top of the white cap tubes will be carefully aspirated using a sterile syringe, while avoiding red blood cells.

The L-PRF clots obtained after 12 minutes of centrifugation will be placed in the Xpression box (IntraSpin, Intra-Lock, Florida, USA) for 5 minutes to allow gentle compression (by gravity) into membranes.

To prepare the L-PRF block, the L-PRF membranes will be cut into small pieces and mixed with the dentin particles at a ratio of 2 membranes to 0.5 g of dentin, providing a 1:1 volume ratio. The liquid fibrinogen will be added to the homogeneous mixture, and while shaping the mixture into the desired form, it will be gently stirred for approximately 10 seconds. Within a few minutes, the fibrinogen will convert into fibrin primarily from the activated blood platelets in the chopped L-PRF membranes. This process will effectively trap the biomaterial and the L-PRF pieces, forming a sturdy block known as the "dentin block," which serves as a convenient and compact graft.

Alveolar ridge preservation: Following a thorough cleaning procedure, the sockets will be carefully packed with customized "dentin blocks" that are shaped to match the individual size and contours of each socket. Once the grafts are properly adapted to the sockets, they will be covered with two layers of L-PRF membranes, which will extend approximately 2 mm along the entire envelope formed between the periosteum and the bony boundaries of the sockets (in a 360° fashion). To ensure stability and prevent displacement, the wounds will be secured using non-resorbable sutures. It's important to note that the purpose of the sutures is to maintain the position of the grafts and membranes rather than closing the wounds entirely.

In the control group: The same extraction and socket debridement procedure will be performed. Following that, the extraction socket will be thoroughly filled with deproteinized bovine bone mineral, and a collagen membrane will be employed to cover the socket. The membrane will be shaped to extend 2-3 mm beyond the margins of the extraction socket and positioned just beneath the marginal mucosa. To ensure its stability, a cross-suture will be performed, securing the membrane in place.

The sutures will be removed two weeks after the surgery.

Biopsy collection: After a healing period of 6 months, at the time of implant placement, a biopsy will be taken from the central area of the grafted site using a 3-mm trephine bur. The biopsy will be promptly fixed in 10% neutral buffered formalin, followed by dehydration through a series of alcohol baths with increasing concentrations (ranging from 50% to 100%). Subsequently, the specimen will be embedded in paraffin. Finally, a tissue section with a thickness of 4 μm will be prepared and subjected to hematoxylin-eosin staining for subsequent histological analysis.

Outcomes: Radiographic vertical buccal bone changes, vertical palatal bone changes, horizontal bone changes, percentage of new vital bone formation, percentage of residual bone graft, and implant primary stability

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-restorable teeth and Type II extraction socket in the esthetic zone
* Healthy patients with adequate oral hygiene (bleeding on probing ≤20%; Plaque index ≤20%).
* Systemically healthy.

Exclusion Criteria:

* Heavy smokers (more than 10 cigarettes per day or an electronic cigarette dose of >6 mg/ml of nicotine).
* Patients reporting systemic conditions that may compromise healing or bone metabolism (eg: diabetes).
* Patients with poor oral hygiene (bleeding on probing >20%; Plaque index >20%)
* The presence of acute periapical infection.
* The presence of severe periodontal destruction.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in radiographic horizontal ridge width | at baseline and 6 months postoperatively
  CBCT scans will be performed at baseline and 6 months postoperatively. Measurements will be taken at both time points using identical reference points and lines. To establish a reference, the most apical point of the extraction socket will be identified on the baseline image, and two reference lines will be drawn. The vertical reference line will be placed at the midpoint of the extraction socket, intersecting the apical reference point. Additionally, a horizontal reference line will be drawn perpendicular to the vertical line, passing through the apical reference point.
  The horizontal ridge width will be measured at three specific levels: 1 mm, 3 mm, and 5 mm below the most coronal aspect of the crest. These measurements will be denoted as HW-1, HW-3, and HW-5, respectively.

SECONDARY OUTCOMES:
Change in radiographic buccal and palatal ridge height | at baseline and 6 months postoperatively
  CBCT scans will be performed at baseline and 6 months postoperatively. Measurements will be taken at both time points using identical reference points and lines. To establish a reference, the most apical point of the extraction socket will be identified on the baseline image, and two reference lines will be drawn. The vertical reference line will be placed at the midpoint of the extraction socket, intersecting the apical reference point.
  The height of the alveolus will be measured at the midbuccal aspect (BH) and midlingual aspect (LH).
Percentage of new vital bone formation and residual graft | after 6 months postoperatively
  The biopsies will be stored in a 10% formalin solution for preservation. Afterward, they will undergo decalcification in EDTA for a duration of four weeks. Following decalcification, the specimens will be processed and embedded in paraffin to create tissue blocks. Longitudinal sections of 5μm thickness will be cut from the paraffin blocks. These sections will be stained using hematoxylin and eosin (H&E) or Masson's trichromatic (MT) stains for histological evaluation and histomorphometric analysis.
Implant Primary Stability | after 6 months postoperatively
  The primary stability of the implant fixture will be assessed using the Osstell Mentor Resonance Frequency Analyzer (Osstell AB, Goteborg, Sweden). Two measurements will be taken in the buccolingual and mesiodistal directions for each implant. The average of these two measurements will be recorded as the representative implant stability quotient (ISQ) for each individual implant.

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hosny, Professor, Study Director — Cairo University
Locations (1):
- Faculty of dentistry Cairo University, Cairo, Elmanil, Egypt